CLINICAL TRIAL: NCT05550662
Title: Hyperpolarized 129Xe Magnetic Resonance Imaging for Evaluation of Chronic Lung Allograft Dysfunction in Lung Transplant Recipients
Brief Title: HP 129Xe MRI for Evaluation of CLAD in Lung Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Giles Santyr, Dr Giles Santyr (PhD), The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1000078240
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Lung Transplant Rejection
Keywords: Lung MRI; 129Xenon; Lung transplant recipient; Chronic lung allograft dysfunction

STUDY DESIGN:
Intervention Model Description: We will map lung ventilation (V), perfusion (Q), apparent diffusion coefficient (ADC) and gas exchange using 129Xe MRI in 15 LTx recipients. All MRI scans will be acquired in one visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Participants will inhale hyperpolarized 129Xe gas.
  Interventions: Drug: 129Xenon

INTERVENTIONS:
Drug: 129Xenon — There is no study medication evaluated. As part of the MRI, participants will inhale hyperpolarized 129Xe gas at a dose of up to 1/6th of total lung capacity (TLC) (lung volume), mixed with nitrogen to a total volume of 1.5 L. The polarized 129Xe will be inhaled in a single breath-hold. This is intended to fill the lungs gas, allowing for lung MRI.
  Other Names: Hyperpolarized Xenon Gas

SUMMARY:
To evaluate the feasibility of hyperpolarized 129Xe MRI in lung transplant recipients and assess structural and functional pulmonary changes using hyperpolarized 129Xe MRI

DETAILED DESCRIPTION:
Lung transplantation is an effective treatment for end-stage lung disease. However, median survival post-LTx is 6 years. This is primarily due to chronic lung allograft dysfunction (CLAD).

Clinical management of LTx recipients is focused on identifying early risk factors for CLAD, by monitoring graft function with spirometry and transbronchial biopsies. However, both have significant limitations.

Hyperpolarized (HP) noble gas lung MRI (3He and 129Xe) allows mapping of both lung anatomy and function. 129Xe-MRI could provide a diagnostic tool that is able to detect CLAD more sensitively and earlier than the current gold standard measurements of spirometry and plethysmography, and thus allow a means to detect and prevent /slow down irreparable and irreversible damage to the lungs in the early stages of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients, deemed clinically stable by the lung transplant team at UHN Toronto Lung Transplant Program (TLTP), 18 years of age or older
* Double lung transplant recipient
* For the 5 CLAD-free participants - at least 1 year of follow-up post-LTx and no substantial and persistent FEV1 decline (as per the ISHLT CLAD definition).
* For the 10 participants with CLAD - prior diagnosis of CLAD made by the clinical team (member of the TLTP).
* PFT measurements within 1 month of scan visit.
* FEV1 > 1.0 L

Exclusion Criteria:

* Currently pregnant or lactating
* Psychiatric or addictive disorders that would preclude obtaining informed consent or adherence to protocol
* Inability to travel to obtain MRI scan
* Any contraindications to MRI including but not limited to severe claustrophobia, implanted devices, aneurysm clips, neurostimulators (patients will be prescreened prior to registration).
* Baseline oxygen saturation of less than 88%.
* Requiring supplemental oxygen at baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
129Xe-MRI | 1 year
  Ventilation defect percent (VDP)

SECONDARY OUTCOMES:
1H-MRI | 1 year
  Structural features

CONTACTS AND LOCATIONS:
Overall Officials: Giles Santyr, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Hospital for Sick Chilldren, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No